CLINICAL TRIAL: NCT05505019
Title: The Role of a Personalized Music Intervention Towards Alleviating Apathy in Parkinson's Disease
Brief Title: Targeting Apathy With Music in Parkinson's Disease
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of British Columbia (Other)
Collaborators: Northeastern University (Other)
Responsible Party: Principal Investigator, Silke Cresswell, Principal Investigator, University of British Columbia
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: H22-00905
Record Dates: First submitted 2022-07-19; First posted 2022-08-17 (Actual); Last update posted 2023-03-17 (Actual); Status verified 2023-03

CONDITIONS: Parkinson Disease; Apathy
Keywords: Music; Music intervention; Non-motor symptoms
MeSH Terms: conditions — Parkinson Disease; Lethargy

STUDY DESIGN:
Intervention Model Description: Participants with Parkinson's Disease (PD) and apathy will be randomly assigned to one of two experimental groups: 1) A music-listening group, and 2) a podcast-listening group.
Who Masked: Participant, Care Provider, Outcomes Assessor
Masking Description: A randomization schedule will be designed by the research coordinator (MJ) and only the research coordinator will know the group allocations. If any experimental condition is shown to be harmful to any participant and it is medically crucial for a participant to know which intervention group they are in, the research coordinator will break code and disclose this information to the participant.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Parkinson's Disease with apathy - Music-listening (Experimental): Participants in this arm will receive a YouTube account app to use. Prior to the start of the intervention, a research team member will guide participants in this group in constructing a playlist of music that they "find rewarding or motivating".
  Interventions: Other: Music listening
- Parkinson's Disease with apathy - Podcast-listening (Experimental): Participants in this arm will receive a YouTube account app to use. Prior to the start of the intervention, a research team member will guide participants in this group in choosing a podcast that they "find rewarding or motivating".
  Interventions: Other: Podcast listening

INTERVENTIONS:
Other: Music listening — This intervention involves listening to participant-selected music that they have evaluated as rewarding/motivating. YouTube Music will be used to build both personalized music and podcast interventions.
  Arms: Parkinson's Disease with apathy - Music-listening
Other: Podcast listening — This intervention involves listening to participant-selected podcasts of neutral content. YouTube Music will be used to build both personalized music and podcast interventions.
  Arms: Parkinson's Disease with apathy - Podcast-listening

SUMMARY:
Parkinson's Disease (PD) is often accompanied by non-motor symptoms that make treatment more difficult. One such symptom is apathy (lack of motivation and emotion). There are no treatments for apathy in PD, and this remains a major unmet need in PD patients. One possible way to target apathy in PD patients is listening to music, which has been shown to help improve apathy in older adults. Little work has explored the mechanism in which music targets apathy. Thus, the goal of this study is to understand how music listening can impact the brain towards decreasing apathy in PD patients.

DETAILED DESCRIPTION:
Apathy is a common neuropsychiatric disturbance that manifests in approximately a quarter of patients in early stages of Parkinson's Disease (PD) and becomes more prevalent over disease progression and cognitive decline. Apathy in PD has been categorized as a distinct behavioural syndrome which can be differentiated from depression and anxiety, and is independently associated with lower functioning in daily life, decreased treatment response, and worse quality of life compared with PD patients without apathy. Characterized by a dysfunction in motivation, or lack of self-initiated goal-directed actions, apathy in PD has been hypothesized to stem from dysfunction in goal-directed reward-seeking networks that rely on dopaminergic transmission in the mesocorticolimbic and frontostriatal pathways, which includes the striatum (includes the nucleus accumbens, or NAc), prefrontal cortex (PFC), hippocampus, and amygdala. Pharmacological trials have attempted to target apathy through the neurotransmitter systems with limited success and sometimes adverse effects. The treatment of apathy remains a major unmet need in PD; thus, it is crucial to develop therapeutic interventions targeting apathy in PD and better understand the underlying mechanisms that may lead to apathy.

Evidence of the positive effects of music-based interventions (MBIs) in both healthy aging and clinical geriatric populations has been examined extensively across the literature. The positive effects of MBIs on alleviating apathy and increasing motivation have been reported in studies focusing on several clinical populations, such as dementia, autism spectrum disorder, and patients undergoing cardiac rehabilitation. A major gap in the MBI clinical trials literature is the lack of attention on the underlying mechanisms in which music can carry out its effects, especially regarding reward pathways. Dysfunction in the reward pathways, which involve the striatum, limbic system, and prefrontal cortices, underlie many disorders, symptoms, and syndromes, and elucidating the role of this underlying network with music is important towards understanding how music can mediate reward deficiencies, such as apathy. Understanding how music works to improve brain functioning is a key gap in understanding how to best inform the development of new therapies and interventions.

Recent work in functional, neurochemical, and pharmacological studies have helped elucidate the role of music in activating reward pathways. Namely, the nucleus accumbens (NAc) has been shown to be involved with processing peak emotionally arousing musical experiences, such as the "chills", and subjective valuations from music. Dopamine transmission in the ventral and dorsal striatum is implicated in regulating this process determined through positron emission tomography (PET) imaging. This work has established the role that the NAc and striatum, and dopaminergic transmission play in processing reward from music and its effects on aspects of cognition, such as motivation, learning, and memory. Thus, the effects of music may be able to mediate the underlying reward system that is compromised in PD patients.

More recently, connectivity between reward and auditory circuits, which include the superior temporal gyrus (STG), superior temporal sulcus (STS) and Heschl's gyrus (HG), have been implicated in musical reward processing and evaluation. No studies to date have observed the immediate and long-term effects of rewarding music on the implicated auditory-reward circuitry and action-oriented behaviour. Thus, this study aims to examine the immediate and longitudinal effects of participant-evaluated rewarding music on clinical apathy measures, connectivity in the auditory-reward networks, and effortful activity in PD patients with and without apathy.

ELIGIBILITY:
Inclusion Criteria:

- Clinical diagnosis of Parkinson's Disease following MDS Parkinson's disease criteria

Exclusion Criteria:

* Participants with atypical Parkinsonism (eg. Progressive supranuclear palsy, multiple system atrophy, drug induced, etc.)
* Epilepsy
* Other neurological disease/complications (eg. myopathy, stroke, brain lesion, MS)
* Significant cognitive impairment (MoCa <21)
* Moderate depression (Beck's Depression Inventory >20)
* Severe/multiple head trauma(s)
* Participants with metal/medical implants, including any of the following: artificial heart valve, brain aneurysm clip, electrical stimulators, ear or eye implant, implanted drug infusion pump, coil, catheter, or filter in any blood vessel, orthopedic hardware such as artificial joint, plate, and/or screws, other metallic prostheses, shrapnel, bullets, or other metal fragments, surgery or tattoos, including tattooed eyeliner, in the last six weeks, cardiac pacemaker, wires or defibrillator, or ferromagnetic aneurysm clip)
* Participants who have gone through specific injuries/brain surgery (eg. an injury where a piece of metal lodged in the eye or orbit)

Ages: 40 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2022-02-09 (Actual); Primary Completion 2023-10-01 (Estimated); Study Completion 2025-10-01 (Estimated)

PRIMARY OUTCOMES:
Change in seed-based functional connectivity between auditory, reward, and motor areas (implicated in musical reward processing) during a music-listening task, before and after an 8-week audio-based intervention | 8 weeks
  fMRI - task-based functional magnetic resonance imaging
Change in seed-based functional connectivity between auditory, reward, and motor areas (implicated in musical reward processing) at rest, before and after an 8-week audio-based intervention | 8 weeks
  rsfMRI - resting state functional magnetic resonance imaging
Change in univariate whole-brain analysis at rest before and after an 8-week audio-based intervention | 8 weeks
  rsfMRI - resting state functional magnetic resonance imaging; observing activity across the brain and in specific regions of interest (ROIs), including reward, auditory, and motor areas
Change in univariate whole-brain analysis during a music listening task before and after an 8-week audio-based intervention | 8 weeks
  fMRI - task-based functional magnetic resonance imaging; observing activity across the brain and in specific regions of interest (ROIs), including reward, auditory, and motor areas
Change in fMRI representational similarity analysis during a music listening task before and after an 8-week audio-based intervention | 8 weeks
  fMRI - task-based functional magnetic resonance imaging; observing correlated BOLD (blood oxygen level dependent) activity across the brain and in specific regions of interest (ROIs), including reward, auditory, and motor areas
Change in fMRI representational similarity analysis at rest before and after an 8-week audio-based intervention | 8 weeks
  rsfMRI - resting state functional magnetic resonance imaging; observing correlated BOLD (blood oxygen level dependent) activity across the brain and in specific regions of interest (ROIs), including reward, auditory, and motor areas
Short-term clinical measure of apathy before and after an 8-week audio-based intervention -Positive and Negative Affective Schedule (PANAS) | 8 weeks
  The PANAS is a self-reported 20-item scale with 2 major subscales: Positive affect score and Negative affect score. Items are scored on a scale of 1-5. Scores range from 10-50 for both the Positive and Negative Affect, with higher scores representing higher levels of Positive/Negative affect.
Short-term clinical measure of apathy after a 4-week washout period post-intervention - Positive and Negative Affective Schedule (PANAS) | 4 weeks
  The PANAS is a self-reported 20-item scale with 2 major subscales: Positive affect score and Negative affect score. Items are scored on a scale of 1-5. Scores range from 10-50 for both the Positive and Negative Affect, with higher scores representing higher levels of Positive/Negative affect.
Short-term clinical measure of apathy before and after an 8-week audio-based intervention - Visual Analogue Scale (VAS) | 8 weeks
  The VAS is a visual scale with a rating from 1-10; participants are to indicate the level of apathy and motivation felt at their current state. Higher values indicate more severe apathy.
Short-term clinical measure of apathy after a 4-week washout period post-intervention - Visual Analogue Scale (VAS) | 4 weeks
  The VAS is a visual scale with a rating from 1-10; participants are to indicate the level of apathy and motivation felt at their current state. Higher values indicate more severe apathy.
Long-term clinical measure of apathy before and after an 8-week audio-based intervention - Starkstein Apathy Scale (SAS) | 8 weeks
  The SAS is a 14-item clinical scale used to evaluate apathy in clinical populations. Higher scores indicate more severe apathy. Scores range from 0-42. Participants who score >=14 are considered as having clinical apathy.
Long-term clinical measure of apathy after a 4-week washout period post-intervention - Starkstein Apathy Scale (SAS) | 4 weeks
  The SAS is a 14-item clinical scale used to evaluate apathy in clinical populations. Higher scores indicate more severe apathy. Scores range from 0-42. Participants who score >=14 are considered as having clinical apathy.
Clinical assessment of apathy before and after an 8-week audio-based intervention - Lille Apathy Rating Scale (LARS) | 8 weeks
  The LARS is a 33-item assessment with 9 subscales: everyday productivity, interests, taking the initiative, novelty seeking, motivation - voluntary actions, emotional responses, concern, social life, and self-awareness. There is a mix of open-ended (items scored between -2 and 2) and multiple choice items (items scored between -1 and 1). Scores range from -36 to 36. Higher scores indicate more severe apathy.
Clinical assessment of apathy after a 4-week washout period post-intervention - Lille Apathy Rating Scale (LARS) | 4 weeks
  The LARS is a 33-item assessment with 9 subscales: everyday productivity, interests, taking the initiative, novelty seeking, motivation - voluntary actions, emotional responses, concern, social life, and self-awareness. There is a mix of open-ended (items scored between -2 and 2) and multiple choice items (items scored between -1 and 1). Scores range from -36 to 36. Higher scores indicate more severe apathy.
Clinical assessment of apathy in Parkinson's Disease before and after an 8-week audio-based intervention - Movement Disorders Society Unified Parkinson's Disease Rating Scale - apathy item (MDS-UPDRS) | 8 weeks
  The MDS-UPDRS is a clinical assessment of motor and non-motor symptoms in individuals with Parkinson's Disease. It consists of four subscales. Subscales 1, 3, and 4 are administered by a trained individual with subscale 2 being self reported. Each item is rated from 0 to 4.
Clinical assessment of apathy in Parkinson's Disease after a 4-week washout period post-intervention - Movement Disorders Society Unified Parkinson's Disease Rating Scale - apathy item | 4 weeks
  The MDS-UPDRS is a clinical assessment of motor and non-motor symptoms in individuals with Parkinson's Disease. It consists of four subscales. Subscales 1, 3, and 4 are administered by a trained individual with subscale 2 being self reported. Each item is rated from 0 to 4.
Assessment of musical reward sensitivity before and after an 8-week audio-based intervention - Barcelona Musical Reward Questionnaire (BMRQ) | 8 weeks
  The BMRQ is a validated 20-item assessment of musical reward sensitivity (how responsive a participant is to the rewarding effects of music listening). It has 5 subscales: musical seeking, emotion evocation, mood regulation, social reward, and sensory-motor. Items are scored from 1-5. Higher scores indicate higher sensitivity to reward.
Assessment of musical reward sensitivity after a 4-week washout period post-intervention - Barcelona Musical Reward Questionnaire (BMRQ) | 4 weeks
  The BMRQ is a validated 20-item assessment of musical reward sensitivity (how responsive a participant is to the rewarding effects of music listening). It has 5 subscales: musical seeking, emotion evocation, mood regulation, social reward, and sensory-motor. Items are scored from 1-5. Higher scores indicate higher sensitivity to reward.
Grip force response (GFR) during a music listening fMRI task before and after an 8-week audio-based intervention | 8 weeks
  GFR is a physical effort measure; it is a validated measure of apathy in Parkinson's Disease (Zhu et al., 2021)
Grip force duration and fatigue during a music listening fMRI task before and after an 8-week audio-based intervention | 8 weeks
  Grip force duration and fatigue are physical effort measures; they are validated measures of apathy in Parkinson's Disease (Zhu et al., 2021)

SECONDARY OUTCOMES:
Clinical assessment for Quality of Life before and after an 8-week audio-based intervention - Quality of Life Scale (QOLS); observing if the intervention improves QoL measures | 8 weeks
  Quality of Life Scale (QOLS)
White and grey matter distribution | 8 weeks
  T1-weighted magnetic resonance image (MRI)

OTHER OUTCOMES:
Clinical assessment for overall cognition - Montreal Cognitive Assessment (MoCA) | 0 weeks (baseline)
  The MoCA is a researcher-administered 30-item assessment covering 8 aspects of cognition: visuospatial/executive, naming, memory, attention, language, abstraction, delayed recall, and orientation. Scores range from 0-30. Higher scores indicate better cognition; lower scores indicate poorer cognition.
Clinical assessment for depressive symptoms (not diagnostic) - Beck's Depression Inventory (BDI) | 0 weeks (baseline)
  The BDI is a self reported 21-question multiple-choice self-report inventory on a scale from 0-3. Scores range from 0-63. Higher scores indicate higher levels of depression; scores over 40 are considered as extreme depression. It will be used as a screening tool to observe any overlap between apathy and depression.
Validated assessment of musical perception (contour subtest) - Montreal Battery of Evaluation of Amusia (MBEA); | 0 weeks (baseline)
  The Montreal Battery of Evaluation of Amusia (MBEA) measures level of general music perception for universal musical structures. This will be used to rule out any non-effects of the music intervention due to a deficit in musical perception abilities; the contour subtest will be used to evaluate this.
Clinical assessment of overall reward/pleasure sensitivity - Snaith-Hamilton Pleasure Scale (SHAPS) | 0 weeks (baseline)
  The SHAPS will be used to compare with BMRQ to isolate for overall anhedonia/apathy versus music-specific apathy (Loui and Belfi, 2020). Higher scores correlate with higher apathy/less pleasure.
White matter tract - axial diffusivity; lesion analysis in white matter tracts (focus on arcuate fasciculus) | 8 weeks
  diffuse tensor image (DTI)
White matter tracts; lesion analysis in white matter tracts (focus on arcuate fasciculus) | 8 weeks
  diffuse tensor image (DTI)

CONTACTS AND LOCATIONS:
Locations (1):
- Djavad Mowafghian Centre for Brain Health, Vancouver, British Columbia, Canada

REFERENCES:
- [Background] Pagonabarraga J, Kulisevsky J. Apathy in Parkinson's Disease. Int Rev Neurobiol. 2017;133:657-678. doi: 10.1016/bs.irn.2017.05.025. Epub 2017 Jul 10. PMID 28802937
- [Background] Pagonabarraga J, Kulisevsky J, Strafella AP, Krack P. Apathy in Parkinson's disease: clinical features, neural substrates, diagnosis, and treatment. Lancet Neurol. 2015 May;14(5):518-31. doi: 10.1016/S1474-4422(15)00019-8. Epub 2015 Apr 12. PMID 25895932
- [Background] Aarsland D, Bronnick K, Alves G, Tysnes OB, Pedersen KF, Ehrt U, Larsen JP. The spectrum of neuropsychiatric symptoms in patients with early untreated Parkinson's disease. J Neurol Neurosurg Psychiatry. 2009 Aug;80(8):928-30. doi: 10.1136/jnnp.2008.166959. PMID 19608786
- [Background] Barone P, Antonini A, Colosimo C, Marconi R, Morgante L, Avarello TP, Bottacchi E, Cannas A, Ceravolo G, Ceravolo R, Cicarelli G, Gaglio RM, Giglia RM, Iemolo F, Manfredi M, Meco G, Nicoletti A, Pederzoli M, Petrone A, Pisani A, Pontieri FE, Quatrale R, Ramat S, Scala R, Volpe G, Zappulla S, Bentivoglio AR, Stocchi F, Trianni G, Dotto PD; PRIAMO study group. The PRIAMO study: A multicenter assessment of nonmotor symptoms and their impact on quality of life in Parkinson's disease. Mov Disord. 2009 Aug 15;24(11):1641-9. doi: 10.1002/mds.22643. PMID 19514014
- [Background] Golebiowski D, van der Bom IMJ, Kwon CS, Miller AD, Petrosky K, Bradbury AM, Maitland S, Kuhn AL, Bishop N, Curran E, Silva N, GuhaSarkar D, Westmoreland SV, Martin DR, Gounis MJ, Asaad WF, Sena-Esteves M. Direct Intracranial Injection of AAVrh8 Encoding Monkey beta-N-Acetylhexosaminidase Causes Neurotoxicity in the Primate Brain. Hum Gene Ther. 2017 Jun;28(6):510-522. doi: 10.1089/hum.2016.109. Epub 2017 Jan 26. PMID 28132521
- [Background] Marin RS. Apathy: Concept, Syndrome, Neural Mechanisms, and Treatment. Semin Clin Neuropsychiatry. 1996 Oct;1(4):304-314. doi: 10.1053/SCNP00100304. PMID 10320433
- [Background] Schmidt L, d'Arc BF, Lafargue G, Galanaud D, Czernecki V, Grabli D, Schupbach M, Hartmann A, Levy R, Dubois B, Pessiglione M. Disconnecting force from money: effects of basal ganglia damage on incentive motivation. Brain. 2008 May;131(Pt 5):1303-10. doi: 10.1093/brain/awn045. Epub 2008 Mar 15. PMID 18344560
- [Background] Chatterjee A, Fahn S. Methylphenidate treats apathy in Parkinson's disease. J Neuropsychiatry Clin Neurosci. 2002 Fall;14(4):461-2. doi: 10.1176/jnp.14.4.461. No abstract available. PMID 12426416
- [Background] Zahodne LB, Bernal-Pacheco O, Bowers D, Ward H, Oyama G, Limotai N, Velez-Lago F, Rodriguez RL, Malaty I, McFarland NR, Okun MS. Are selective serotonin reuptake inhibitors associated with greater apathy in Parkinson's disease? J Neuropsychiatry Clin Neurosci. 2012 Summer;24(3):326-30. doi: 10.1176/appi.neuropsych.11090210. PMID 23037646
- [Background] Lam HL, Li WTV, Laher I, Wong RY. Effects of Music Therapy on Patients with Dementia-A Systematic Review. Geriatrics (Basel). 2020 Sep 25;5(4):62. doi: 10.3390/geriatrics5040062. PMID 32992767
- [Background] Tsoi KKF, Chan JYC, Ng YM, Lee MMY, Kwok TCY, Wong SYS. Receptive Music Therapy Is More Effective than Interactive Music Therapy to Relieve Behavioral and Psychological Symptoms of Dementia: A Systematic Review and Meta-Analysis. J Am Med Dir Assoc. 2018 Jul;19(7):568-576.e3. doi: 10.1016/j.jamda.2017.12.009. Epub 2018 Feb 1. PMID 29396186
- [Background] Tang Q, Zhou Y, Yang S, Thomas WKS, Smith GD, Yang Z, Yuan L, Chung JW. Effect of music intervention on apathy in nursing home residents with dementia. Geriatr Nurs. 2018 Jul-Aug;39(4):471-476. doi: 10.1016/j.gerinurse.2018.02.003. Epub 2018 Mar 15. PMID 29551546
- [Background] Goris ED, Ansel KN, Schutte DL. Quantitative systematic review of the effects of non-pharmacological interventions on reducing apathy in persons with dementia. J Adv Nurs. 2016 Nov;72(11):2612-2628. doi: 10.1111/jan.13026. Epub 2016 Jun 23. PMID 27221007
- [Background] Quintin EM. Music-Evoked Reward and Emotion: Relative Strengths and Response to Intervention of People With ASD. Front Neural Circuits. 2019 Sep 18;13:49. doi: 10.3389/fncir.2019.00049. eCollection 2019. PMID 31619969
- [Background] Bowles L, Curtis J, Davies C, Lengerich A, Bugajski A. The effect of music on mood, motivation, and exercise among patients in a cardiac rehabilitation program: A pilot study. Nurs Forum. 2019 Jul;54(3):340-344. doi: 10.1111/nuf.12334. Epub 2019 Feb 25. PMID 30802308
- [Background] Le Heron C, Holroyd CB, Salamone J, Husain M. Brain mechanisms underlying apathy. J Neurol Neurosurg Psychiatry. 2019 Mar;90(3):302-312. doi: 10.1136/jnnp-2018-318265. Epub 2018 Oct 26. PMID 30366958
- [Background] Volkow ND, Michaelides M, Baler R. The Neuroscience of Drug Reward and Addiction. Physiol Rev. 2019 Oct 1;99(4):2115-2140. doi: 10.1152/physrev.00014.2018. PMID 31507244
- [Background] Adam TC, Epel ES. Stress, eating and the reward system. Physiol Behav. 2007 Jul 24;91(4):449-58. doi: 10.1016/j.physbeh.2007.04.011. Epub 2007 Apr 14. PMID 17543357
- [Background] Martin-Soelch C. Is depression associated with dysfunction of the central reward system? Biochem Soc Trans. 2009 Feb;37(Pt 1):313-7. doi: 10.1042/BST0370313. PMID 19143654
- [Background] Salimpoor VN, Benovoy M, Larcher K, Dagher A, Zatorre RJ. Anatomically distinct dopamine release during anticipation and experience of peak emotion to music. Nat Neurosci. 2011 Feb;14(2):257-62. doi: 10.1038/nn.2726. Epub 2011 Jan 9. PMID 21217764
- [Background] Blood AJ, Zatorre RJ. Intensely pleasurable responses to music correlate with activity in brain regions implicated in reward and emotion. Proc Natl Acad Sci U S A. 2001 Sep 25;98(20):11818-23. doi: 10.1073/pnas.191355898. PMID 11573015
- [Background] Gold BP, Mas-Herrero E, Zeighami Y, Benovoy M, Dagher A, Zatorre RJ. Musical reward prediction errors engage the nucleus accumbens and motivate learning. Proc Natl Acad Sci U S A. 2019 Feb 19;116(8):3310-3315. doi: 10.1073/pnas.1809855116. Epub 2019 Feb 6. PMID 30728301
- [Background] Menon V, Levitin DJ. The rewards of music listening: response and physiological connectivity of the mesolimbic system. Neuroimage. 2005 Oct 15;28(1):175-84. doi: 10.1016/j.neuroimage.2005.05.053. Epub 2005 Jul 14. PMID 16023376
- [Background] Ferreri L, Mas-Herrero E, Zatorre RJ, Ripolles P, Gomez-Andres A, Alicart H, Olive G, Marco-Pallares J, Antonijoan RM, Valle M, Riba J, Rodriguez-Fornells A. Dopamine modulates the reward experiences elicited by music. Proc Natl Acad Sci U S A. 2019 Feb 26;116(9):3793-3798. doi: 10.1073/pnas.1811878116. Epub 2019 Jan 22. PMID 30670642
- [Background] Ferreri L, Mas-Herrero E, Cardona G, Zatorre RJ, Antonijoan RM, Valle M, Riba J, Ripolles P, Rodriguez-Fornells A. Dopamine modulations of reward-driven music memory consolidation. Ann N Y Acad Sci. 2021 Oct;1502(1):85-98. doi: 10.1111/nyas.14656. Epub 2021 Jul 11. PMID 34247392
- [Background] Salimpoor VN, van den Bosch I, Kovacevic N, McIntosh AR, Dagher A, Zatorre RJ. Interactions between the nucleus accumbens and auditory cortices predict music reward value. Science. 2013 Apr 12;340(6129):216-9. doi: 10.1126/science.1231059. PMID 23580531
- [Background] Belfi AM, Loui P. Musical anhedonia and rewards of music listening: current advances and a proposed model. Ann N Y Acad Sci. 2020 Mar;1464(1):99-114. doi: 10.1111/nyas.14241. Epub 2019 Sep 23. PMID 31549425
- [Background] Zatorre RJ. Why Do We Love Music? Cerebrum. 2018 Nov 1;2018:cer-16-18. eCollection 2018 Nov-Dec. PMID 30746026
- [Background] Berridge KC, Kringelbach ML. Affective neuroscience of pleasure: reward in humans and animals. Psychopharmacology (Berl). 2008 Aug;199(3):457-80. doi: 10.1007/s00213-008-1099-6. Epub 2008 Mar 3. PMID 18311558
- [Background] Berridge KC, Robinson TE. Liking, wanting, and the incentive-sensitization theory of addiction. Am Psychol. 2016 Nov;71(8):670-679. doi: 10.1037/amp0000059. PMID 27977239
- [Background] Husain M, Roiser JP. Neuroscience of apathy and anhedonia: a transdiagnostic approach. Nat Rev Neurosci. 2018 Aug;19(8):470-484. doi: 10.1038/s41583-018-0029-9. PMID 29946157
- [Background] Ducharme S, Price BH, Dickerson BC. Apathy: a neurocircuitry model based on frontotemporal dementia. J Neurol Neurosurg Psychiatry. 2018 Apr;89(4):389-396. doi: 10.1136/jnnp-2017-316277. Epub 2017 Oct 24. PMID 29066518
- [Background] Salimpoor VN, Benovoy M, Longo G, Cooperstock JR, Zatorre RJ. The rewarding aspects of music listening are related to degree of emotional arousal. PLoS One. 2009 Oct 16;4(10):e7487. doi: 10.1371/journal.pone.0007487. PMID 19834599
- [Background] Yang M, He H, Duan M, Chen X, Chang X, Lai Y, Li J, Liu T, Luo C, Yao D. The Effects of Music Intervention on Functional Connectivity Strength of the Brain in Schizophrenia. Neural Plast. 2018 May 2;2018:2821832. doi: 10.1155/2018/2821832. eCollection 2018. PMID 29853841
- [Background] Starkstein SE, Mayberg HS, Preziosi TJ, Andrezejewski P, Leiguarda R, Robinson RG. Reliability, validity, and clinical correlates of apathy in Parkinson's disease. J Neuropsychiatry Clin Neurosci. 1992 Spring;4(2):134-9. doi: 10.1176/jnp.4.2.134. PMID 1627973
- [Background] Watson D, Clark LA, Tellegen A. Development and validation of brief measures of positive and negative affect: the PANAS scales. J Pers Soc Psychol. 1988 Jun;54(6):1063-70. doi: 10.1037//0022-3514.54.6.1063. PMID 3397865
- [Background] Tinaz S, Kamel S, Aravala SS, Sezgin M, Elfil M, Sinha R. Distinct neural circuits are associated with subclinical neuropsychiatric symptoms in Parkinson's disease. J Neurol Sci. 2021 Apr 15;423:117365. doi: 10.1016/j.jns.2021.117365. Epub 2021 Feb 21. PMID 33636663
- [Background] Smith CR, Cavanagh J, Sheridan M, Grosset KA, Cullen B, Grosset DG. Factor structure of the Montreal Cognitive Assessment in Parkinson disease. Int J Geriatr Psychiatry. 2020 Feb;35(2):188-194. doi: 10.1002/gps.5234. Epub 2019 Dec 3. PMID 31736141
- [Background] Richter P, Werner J, Heerlein A, Kraus A, Sauer H. On the validity of the Beck Depression Inventory. A review. Psychopathology. 1998;31(3):160-8. doi: 10.1159/000066239. PMID 9636945
- [Background] Snaith RP, Hamilton M, Morley S, Humayan A, Hargreaves D, Trigwell P. A scale for the assessment of hedonic tone the Snaith-Hamilton Pleasure Scale. Br J Psychiatry. 1995 Jul;167(1):99-103. doi: 10.1192/bjp.167.1.99. PMID 7551619
- [Background] Nunes-Silva M, Haase VG. Montreal Battery of Evaluation of Amusia: Validity evidence and norms for adolescents in Belo Horizonte, Minas Gerais, Brazil. Dement Neuropsychol. 2012 Oct-Dec;6(4):244-252. doi: 10.1590/S1980-57642012DN06040008. PMID 29213804
- [Background] Burckhardt CS, Anderson KL. The Quality of Life Scale (QOLS): reliability, validity, and utilization. Health Qual Life Outcomes. 2003 Oct 23;1:60. doi: 10.1186/1477-7525-1-60. PMID 14613562
- [Background] Zhang Y, Zhang GY, Zhang ZE, He AQ, Gan J, Liu Z. White matter hyperintensities: a marker for apathy in Parkinson's disease without dementia? Ann Clin Transl Neurol. 2020 Sep;7(9):1692-1701. doi: 10.1002/acn3.51159. Epub 2020 Aug 28. PMID 32857484
- [Background] Martinez-Molina N, Mas-Herrero E, Rodriguez-Fornells A, Zatorre RJ, Marco-Pallares J. White Matter Microstructure Reflects Individual Differences in Music Reward Sensitivity. J Neurosci. 2019 Jun 19;39(25):5018-5027. doi: 10.1523/JNEUROSCI.2020-18.2019. Epub 2019 Apr 18. PMID 31000588
- [Background] Loui P, Patterson S, Sachs ME, Leung Y, Zeng T, Przysinda E. White Matter Correlates of Musical Anhedonia: Implications for Evolution of Music. Front Psychol. 2017 Sep 25;8:1664. doi: 10.3389/fpsyg.2017.01664. eCollection 2017. PMID 28993748
- [Background] Chomiak T, Watts A, Meyer N, Pereira FV, Hu B. A training approach to improve stepping automaticity while dual-tasking in Parkinson's disease: A prospective pilot study. Medicine (Baltimore). 2017 Feb;96(5):e5934. doi: 10.1097/MD.0000000000005934. PMID 28151878
- [Background] Zhu M, HajiHosseini A, Baumeister TR, Garg S, Appel-Cresswell S, McKeown MJ. Altered EEG alpha and theta oscillations characterize apathy in Parkinson's disease during incentivized movement. Neuroimage Clin. 2019;23:101922. doi: 10.1016/j.nicl.2019.101922. Epub 2019 Jul 2. PMID 31284232